CLINICAL TRIAL: NCT01179971
Title: Incorporation of n-3 Long Chain Polyunsaturated Fatty Acids and Gamma Linolenic Acid in Plasma Lipids, Cholesteryl Esters, and Erythrocyte Membranes and Their Influence on Disease Activity in Patients With Rheumatoid Arthritis
Brief Title: n-3 and n-6 Fatty Acids in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Jena (Other)
Responsible Party: Rainer Stange, M.D. Ph.D., Abteilung für Naturheilkunde Charité
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Charite-n-3-n-6
Record Dates: First submitted 2010-08-04; First posted 2010-08-11 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Rheumatoid Arthritis
Keywords: n-3 fatty acids; n-6 fatty acids; anti-inflammatory action; clinical trial; randomized double-blinded; incorporation of fatty acids
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Fish Oils; gamma-Linolenic Acid; Fatty Acids, Omega-6

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fish oil (Experimental): 3g/d
  Interventions: Dietary Supplement: Fish oil, gamma-linolenic acid
- Gamma-linolenic Acid (Experimental): 3g/d gamma-linolenic acid
  Interventions: Dietary Supplement: Fish oil, gamma-linolenic acid
- Fish oil plus GLA (Experimental): 1.5 g/d DHA + EPA plus 1.5g/d gamma-linolenic acid
  Interventions: Dietary Supplement: Fish oil, gamma-linolenic acid
- Olive oil (Sham Comparator): 3 g/d olive oil
  Interventions: Dietary Supplement: Fish oil, gamma-linolenic acid

INTERVENTIONS:
Dietary Supplement: Fish oil, gamma-linolenic acid — 3 g/d DHA + EPA
  Other Names: Fish oil, omega-6 fatty acids

SUMMARY:
Purpose: To investigate into the differential effects of polyunsaturated fatty acids as compared to standard control therapy (olive oil) on disease activity and biochemical parameters in patients with rheumatoid arthritis (RA), resp. psoriasis arthritis (PA).

DETAILED DESCRIPTION:
Methods: Double-blinded, four-armed randomised controlled trial with 3.0 g/d of either n-3 long chain polyunsaturated fatty acids (LC-PUFA) or gamma linolenic acid (GLA), resp. the combination of 1.5 g/d of each, resp. 3.0 g/d of olive oil over 12 weeks. Outcome parameters disease activity score (DAS28), C-reactive protein, concentrations of n-3 LC-PUFA, resp. GLA in plasma lipids (PL), cholesterol esters (CE), and erythrocyte membranes (EM), and serum concentrations of arachidonic acid (AA). Conventional antirheumatic and immunosuppressive therapies could be changed only within defined limits.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid or Psoriasis arthritis

Exclusion Criteria:

* Severe diseases of heart, liver, lung airways
* Non-compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
incorporation of eicosapentaenoic acid in plasma lipids | 12 weeks
  ratio of arachidonic acid/eicosapentaenoic acid in plasma lipids

SECONDARY OUTCOMES:
Disease activity score 28 (DAS28, EULAR) | 12 weeks
  Disease activity as determinated by counts of swollen and tender joints, patient's judgement and erythrocyte sedimentation rate
C-reactive protein | 12 weeks
  most common marker of acute systemic inflammation
International Normalized Ratio (INR) | 12 weeks
  most common single marker for crude quantification of hemostasis
Tolerability | 12 weeks
  registration of complaints for taste, odor, or mechanical properties of the supplements

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Stange, MD, PhD, Principal Investigator — Immanuel Krankenhaus and Charite Berlin

REFERENCES:
- [Derived] Dawczynski C, Hackermeier U, Viehweger M, Stange R, Springer M, Jahreis G. Incorporation of n-3 PUFA and gamma-linolenic acid in blood lipids and red blood cell lipids together with their influence on disease activity in patients with chronic inflammatory arthritis--a randomized controlled human intervention trial. Lipids Health Dis. 2011 Aug 4;10:130. doi: 10.1186/1476-511X-10-130. PMID 21816071